CLINICAL TRIAL: NCT06566170
Title: Long-Term Real-World Comparative Effectiveness of Donanemab Plus Usual Care Versus Usual Care Alone in US Patients With Early Symptomatic Alzheimer's Disease (TRAILBLAZER-REAL US)
Brief Title: A Real-World Comparative Study of Donanemab (LY3002813) Plus Usual Care Versus Usual Care Alone in US Participants With Early Symptomatic Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 18721; I5T-MC-AACS (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — donanemab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Donanemab Group + Usual Care: Participants will receive open-label (unblinded) donanemab intravenously (IV) and Usual Care
  Interventions: Drug: Donanemab; Drug: Usual Care
- Usual Care Group: Participants will receive usual care.
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: Donanemab — Administered IV
  Other Names: LY3002813
  Groups: Donanemab Group + Usual Care
Drug: Usual Care — Medication (excluding amyloid-targeting agents) or non-pharmacological therapy including watchful waiting.

SUMMARY:
The main purpose of this study is to evaluate the long-term effectiveness of donanemab plus usual care versus usual care alone in participants with early symptomatic AD. The study will employ a prospective, observational cohort design with participant management resembling real-world practice to the greatest extent possible via prospective assessments and linkage to historical and prospective electronic health records. The study will last about 273 weeks and may include up to 28 visits.

ELIGIBILITY:
Inclusion Criteria:

Participants

* are under care for presumed mild cognitive impairment (MCI) or mild dementia stage of AD (Note: neither a biomarker-based diagnosis of AD nor a diagnosis in electronic health records [EHR] is required prior to screening)
* have a Telephone Interview for Cognitive Status (TICS) score of ≥21
* presence of amyloid beta (Aβ) pathology supported by biomarker results (e.g., P-tau, amyloid positron emission tomography (PET), and/or cerebrospinal fluid [CSF]). (Note: A historical biomarker may be used for eligibility if performed within 12 months of study entry)
* have a reliable study partner who is in frequent contact with the participant and will be available by telephone at designated times (every 6 months), and
* have EHR data available for linkage and are willing to allow access to EHR data for the duration of the study.

Exclusion Criteria:

* have prior ischemic or hemorrhagic stroke(s) with an inability to independently perform any one or more basic activities of daily living (ADLs) (i.e., walking, transferring, eating, bathing, dressing, or toileting). (Note: mixed dementias with amyloid pathology are permitted)
* have current or recent serious or unstable illness (other than AD) that, in the investigator's opinion, could interfere with the ability of the participant or study partner to complete the study (e.g., life expectancy of less than 36 months, requirement for long-term (>12 months) institutional-level care, serious psychiatric illness, etc.)
* are currently enrolled or intend to enroll in a clinical trial of another investigational product, and
* have contraindications to donanemab, magnetic resonance imaging (MRI), or amyloid PET tracers. (Donanemab group only).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a donanemab plus usual care group and a usual care alone group. Participants will be enrolled 1:2 into donanemab plus usual care and usual care alone groups to allow enough participants in the usual care group to be matched with participants in the donanemab group to enable robust comparative effectiveness analyses.
Sampling Method: Non-Probability Sample
Enrollment: 6250 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2033-02 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Time to First Increase in Dependence Level Above Baseline (as derived from the Dependence Scale [DS]) | Up to 5 Years
  The DS is a caregiver-reported outcome assessing the need for daily in-home or institutional assistance by participants with AD. The DS is completed as a structured interview with a knowledgeable caregiver or study partner. The scale is composed of 13 items evaluating progressive needs for assistance. The total score ranges from 0 to 15, with higher scores indicating a greater degree of dependence on external support.

SECONDARY OUTCOMES:
Time to Loss of Independence (Dependence Level ≥3 as derived from the DS) for the Subgroup of Participants with Dependence Level <3 at Baseline | Up to 5 Years
Time to Institutionalization from Baseline for the Subgroup of Participants not Institutionalized at Baseline | Up to 5 Years
  Participants who endorse, "Assisted living facility" or "Skilled nursing facility, nursing home, hospice" as their primary residence on the participant lifestyle status Questionnaire (P-LSQ) will be considered institutionalized.
Change from Baseline Over Time (Semi-Annually) in DS Total Score | Baseline, Up to 5 Years
Change from Baseline Over Time (Assessed Semi-Annually) in Functional Assessment Questionnaire (FAQ) Total Score | Baseline, Up to 5 Years
  The FAQ is a brief, 10-item caregiver-reported outcome measure assessing performance on functional activities impacted early during AD. The maximum total score is 30, with higher scores indicating greater impairment.
Change from Baseline Over Time (Assessed Yearly) in Neuropsychiatric Inventory (NPI-Q) Total Severity Score | Baseline, Up to 5 Years
  The NPI-Q is a brief, caregiver-reported assessment of neuropsychiatric symptoms associated with dementia. The NPI-Q yields total scores for Severity and Distress, reflecting the sum of ratings across all domains, with higher scores indicating a greater degree of symptom severity and caregiver distress, respectively.
Change from Baseline Over Time (Assessed Yearly) in Zarit Burden Inventory-short version (ZBI-12) total score | Baseline, Up to 5 Years
  ZBI is a caregiver-reported instrument used widely to evaluate caregiver burden associated with AD and other diseases such as multiple sclerosis, congestive heart failure, and cancer. Items on the ZBI-12 assess caregiver stress, time available for self, and the impact of caring on the caregiver's social life. Responses are provided on a 5-point Likert scale (never=0, nearly always=4). The ZBI-12 total score has a range of 0 to 48, with higher scores indicating greater caregiver burden.
Change from Baseline Over Time (Assessed Semi-Annually) in Living Situation as Assessed by the Participant Lifestyle Questionnaire (P-LSQ) | Baseline, Up to 5 Years
  The P-LSQ is a brief, sponsor-created questionnaire used to collect supplementary data regarding participants' living environment, home healthcare needs, and driving status that is not captured elsewhere.
Change from Baseline Over Time (Assessed Semi-Annually) in Home Healthcare as Assessed by the P-LSQ | Baseline, Up to 5 Years
Change from Baseline Over Time (Assessed Semi-Annually) in Driving Status as Assessed by the P-LSQ | Baseline, Up to 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Rehabilitation & Neurological Services, Huntsville, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
URL: http://vivli.org/